CLINICAL TRIAL: NCT02541448
Title: A Single Center, Prospective, Randomized, Controlled Study To Evaluate Physician Preference Related to the Use of the SURGIQUEST AIRSEAL® INSUFFLATION SYSTEM (AIS) at Low VS. Higher Pressure for the Management of Pneumoperitoneum.
Brief Title: Pneumoperitoneum Management With SurgiQuest AirSeal at Low vs. Higher Pressure ( PRESSURE )
Acronym: PRESSURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cynthia Harris (Industry)
Collaborators: SurgiQuest, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Cynthia Harris, Director of Clinical Studies, SurgiQuest, Inc.
Organization: SurgiQuest, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRT DD030316
Record Dates: First submitted 2015-09-01; First posted 2015-09-04 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AIS at 9±1mmHg (Active Comparator): Use of the SurgiQuest AIRSEAL® Insufflation System (AIS) at 9±1mmHg
  Interventions: Device: SurgiQuest AIRSEAL® Insufflation System (AIS)
- AIS at 15±1mmHg (Active Comparator): Use of the SurgiQuest AIRSEAL® Insufflation System (AIS) at 15±1mmHg.
  Interventions: Device: SurgiQuest AIRSEAL® Insufflation System (AIS)

INTERVENTIONS:
Device: SurgiQuest AIRSEAL® Insufflation System (AIS) — The SurgiQuest AirSeal Optical Trocar & Cannula System with integrated Insufflator DPIS 2000 (the "DPIS 2000 System") is intended for use in diagnostic and/or therapeutic endoscopic procedures to distend the peritoneal cavity by filling it with gas (establish and maintain pneumoperitoneum), to establish and maintain a path of entry for endoscopic instruments, and to evacuate surgical smoke. The trocar of the DPIS 2000 System is indicated for use with or without visualization.
  Other Names: AIS

SUMMARY:
This study is designed to evaluate physician preference related to the use of the SURGIQUEST AIRSEAL® INSUFFLATION SYSTEM (AIS) at low verses high pressure for the management of pneumoperitoneum.

DETAILED DESCRIPTION:
The objective of this study is to evaluate physician preferences related to use of the SurgiQuest AirSeal Insufflation System (AIS) used at low vs. higher pressures for maintaining pneumoperitoneum during laparoscopic/robotic surgical procedures.

The study is designed and powered to demonstrate superiority of the AIS used at low insufflation pressure (9±mmHg ±1mmHg) vs higher pressure (15mmHg ±1mmHg) in relation to a single key effectiveness measure: Incidence of shoulder pain. Patients will be randomized 1:1 to either AIS with an insufflation pressure target of 9±1mmHg) or to AIS with an insufflation target pressure of 15±1mmHg.

Secondary outcome measures include severity of shoulder pain measured using a VAS scale and medication use, procedure time, the number of procedure interruptions, length of hospital stay, aspects of anesthesia management including end tidal CO2 and the frequency of adverse events. These outcomes will be evaluated in a controlled population undergoing laparoscopic/robotic surgery.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 80 years of age;
2. Capable and willing to give informed consent;
3. Acceptable candidate for an elective, non-emergent laparoscopic/robotic surgery;

Exclusion Criteria:

1. Advanced refusal of blood transfusion, if necessary;
2. Active systemic or cutaneous infection or inflammation;
3. Pre-existing immunodeficiency disorder and/or chronic use of systemic steroids;
4. Uncontrolled diabetes mellitus
5. Known, significant history of bleeding diathesis, coagulopathy, Von Willebrand's disease or current platelet count < 100,000 cells/mm3, baseline INR ≥1.8, or fibrinogen level less than 150 mg/dl (if received a fibrinolytic agent within prior 24 hours);
6. Severe co-existing morbidities having a life expectancy of less than 30 days;
7. Currently involved in any other investigational clinical Studies;
8. Significant anemia with a hemoglobin level less than 10 g/dL or a hematocrit less than 30%;
9. Renal insufficiency (serum creatinine of > 2.5 mg/dl);
10. Females who are pregnant, planning to become pregnant within 3 months of the procedure, or lactating;
11. Extreme morbid obesity (BMI greater than 45 kg/m2) or underweight (BMI less than 20 kg/m2);
12. Patients presenting with Ascites -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-05-18 (Actual); Study Completion 2018-07-12 (Actual)

PRIMARY OUTCOMES:
Incidence of shoulder pain | participants will be followed for the duration of hospital stay, an expected average of 24 hours
  Incidence of reported shoulder pain

CONTACTS AND LOCATIONS:
Overall Officials: John P Diaz, MD, Principal Investigator — South Miami Hospital, Miami Floridaa
Locations (1):
- South Miami Hospital, Miami, Florida, United States